CLINICAL TRIAL: NCT03852797
Title: Spontaneous and Oxytocin-induced Contractility After Exposure to Intravenous Anesthetic Agents: an In-vitro Study in Human Myometrium
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-01
Record Dates: First submitted 2019-02-21; First posted 2019-02-25 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Postpartum Hemorrhage
Keywords: uterine contraction; oxytocin; ketamine; propofol; etomidate
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Oxytocin; Ketamine; Propofol; Etomidate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Ketamine (Active Comparator): The myometrial samples are bathed in physiological salt solution (PSS) with increasing concentrations of ketamine (from 10 -7M to 10 -4M)
  Interventions: Drug: Ketamine
- Ketamine + oytocin (Active Comparator): The myometrial samples are bathed in an oxytocin solution (20nM) with increasing concentrations of ketamine (from 10 -7M to 10 -4M)
  Interventions: Drug: Oxytocin; Drug: Ketamine
- Propofol (Active Comparator): The myometrial samples are bathed in physiological salt solution (PSS) with increasing concentrations of propofol (from 10 -7M to 10 -4M)
  Interventions: Drug: Propofol
- Propofol + oytocin (Active Comparator): The myometrial samples are bathed in an oxytocin solution (20nM) with increasing concentrations of propofol (from 10 -7M to 10 -4M)
  Interventions: Drug: Oxytocin; Drug: Propofol
- Etomidate (Active Comparator): The myometrial samples are bathed in physiological salt solution (PSS) with increasing concentrations of etomidate (from 10 -7M to 10 -4M)
  Interventions: Drug: Etomidate
- Etomidate + oytocin (Active Comparator): The myometrial samples are bathed in an oxytocin solution (20nM) with increasing concentrations of etomidate (from 10 -7M to 10 -4M)
  Interventions: Drug: Oxytocin; Drug: Etomidate

INTERVENTIONS:
Drug: Oxytocin — Oxytocin solution, 20nM concentration
  Other Names: pitocin
  Arms: Etomidate + oytocin; Ketamine + oytocin; Propofol + oytocin
Drug: Ketamine — Ketamine in solution, 10-4M to 10-7M
  Other Names: ketamine HCl
  Arms: Ketamine; Ketamine + oytocin
Drug: Propofol — Propofol in solution, 10-4M to 10-7M
  Arms: Propofol; Propofol + oytocin
Drug: Etomidate — Etomidate in solution, 10-4M to 10-7M
  Arms: Etomidate; Etomidate + oytocin

SUMMARY:
Poor uterine tone after the birth of a baby may cause serious bleeding (called postpartum hemorrhage or PPH). This is a major cause of maternal death worldwide. In the developed world the cesarean section rate is increasing. There are two modalities for anesthesia for cesarean section; general and regional (eg. spinal anesthetic). General anesthesia has been associated with increased blood loss compared to regional and the reasons for this may be multifactorial. Some of the anesthesia gases have been studied and there is laboratory evidence to suggest that these gases may reduce the tone of the uterus and therefore cause increased blood loss due to poor uterine tone. To date there has been little study on the intravenous anesthesia agents. These agents are usually administered to anaesthetise the patient at the start of surgery (induction of anesthesia), however they can also be used instead of the gases to keep the patient asleep using a 'total intravenous anesthesia' technique. Laboratory work in rats has suggested that high doses of these intravenous drugs might reduce uterine tone, thus increasing the risk of blood loss. Interestingly, at low doses one of these drugs (ketamine) may actually increase uterine tone. Only one of these drugs has been studied in human uterine tissue. The investigators plan to compare three anaesthesia induction agents on human uterine tissue under physiological conditions in the laboratory.

This study will be the first to compare these three drugs on human tissue. The investigators plan to determine the impact of these drugs on spontaneous uterine contractility and also contractilty induced by oxytocin, which is the drug most commonly administered to help contract the uterus after birth. This is important as it will help inform anesthesiologists as to the best drug to use depending on the clinical circumstance.

The investigators hypothesize that the intravenous induction agents will cause a dose dependent decrease in spontaneous uterine contractility, similar to what has been described in the rat model. The investigators also expect that exposure to high concentrations of intravenous anesthesia induction agents will cause a blunted contractile response to oxytocin.

DETAILED DESCRIPTION:
There is an increasing need to fully understand the mechanisms that contribute to the higher blood loss after general anesthesia during cesarean section therefore it is important the investigators identify all pharmacological contributors to poor uterine tone. Furthermore, anesthesiologists are increasingly called upon to care for women undergoing a range of in-utero fetal surgeries which require a careful balanced anesthetic and strict control of uterine tone.

This will be the first study that compares the three commonly used intravenous anesthesia agents on human myometrium: ketamine, etomidate and propofol. This study is required to allow doctors make informed decisions about which anesthesia agent is most suitable to manage their patient depending on clinical circumstances.

The specific objective of this project is to investigate the pharmacological dose-response profiles of different anesthesia induction agents by in-vitro isometric tension measurements of contractions in gravid human myometrium. The investigators will study both spontaneous and oxytocin induced contractility.

ELIGIBILITY:
Inclusion Criteria:

* Patients who give written consent to participate in this study
* Patients with gestational age 37-41 weeks
* Patients of 19-50 years
* Non-laboring patients, not exposed to exogenous oxytocin
* Patients requiring primary Cesarean section or first repeat Cesarean section
* Patients undergoing Cesarean section under spinal anesthesia

Exclusion Criteria:

* Patients who refuse to give written informed consent
* Patients who require general anesthesia
* Patients who had previous uterine surgery or more than one previous Cesarean section
* Patients with any condition predisposing to uterine atony and postpartum hemorrhage, such as abnormal placentation, multiple gestation, preeclampsia, macrosomia, polyhydramnios, uterine fibroids, bleeding diathesis, chorioamnionitis, or a previous history of postpartum bleeding
* Emergency Cesarean section in labor
* Patients on medications that could affect myometrial contractility, such as nifedipine, labetolol or magnesium sulphate.
* Patients who have been exposed to oxytocin prior or during the cesarean section.

Ages: 19 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2019-03-28 (Actual); Primary Completion 2022-01-19 (Actual); Study Completion 2022-01-19 (Actual)

PRIMARY OUTCOMES:
Motility index | 4 hours
  Motility index (MI) is a calculated outcome, based on the formula: frequency/(10 x amplitude).
  Frequency and amplitude are secondary outcome measures as described below.
  The analysis is undertaken by attaching myometrial strips between an isometric force transducer and the base of an organ bath chamber.

SECONDARY OUTCOMES:
Amplitude of contraction | 4 hours
  The maximum extent of uterine muscle contraction, measured in grams (g). The analysis is undertaken by attaching myometrial strips between an isometric force transducer and the base of an organ bath chamber.
Frequency of contraction | 4 hours
  The number of contractions in uterine muscle (myometrium) over 10 minutes, spontaneously and in response to an agonist.
  The analysis is undertaken by attaching myometrial strips between an isometric force transducer and the base of an organ bath chamber.
Integrated area under response curve (AUC) | 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Mrinalini Balki, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada